CLINICAL TRIAL: NCT02618278
Title: Physiotherapy Management of Lumbar Radicular Syndrome; Does Early Intervention Improve Outcomes?
Brief Title: Physiotherapy for Sciatica; Is Earlier Better?
Acronym: POLAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Michael Reddington (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor-Investigator, Michael Reddington, NIHR Clinical Doctoral Research Fellow, Sheffield Teaching Hospitals NHS Foundation Trust
Organization: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STH18420
Record Dates: First submitted 2015-11-23; First posted 2015-12-01 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Sciatica; Low Back Pain; Radiculopathy
MeSH Terms: conditions — Sciatica; Low Back Pain; Radiculopathy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Patients randomised to the intervention arm will receive a individual, goal -orientated physiotherapy management package within 2 weeks G.P referral for physiotherapy.
  Interventions: Other: Physiotherapy
- Usual care (Active Comparator): Patients randomised to usual care will receive the same individual, goal-orientated physiotherapy management as the intervention arm but at 6 weeks post G.P referral, as is usual care.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — The aims of physiotherapy are to promote physical and psychological health for the patient, and in doing so promote and improve function. In light of the evidence to suggest spontaneous resorption of the disc fragment occurs, physiotherapy provides support and guidance for the patient to manage their symptoms whilst resorption takes place. The physiotherapy regimen will be tailored to the individuals' requirements. It will be goal orientated, and assessed using a biopsychosocial approach based on 7 different elements; neurological dysfunction, motor control of movement of the lumbar spine and pelvis, movement restriction in the lumbar spine and pelvis, psychological barriers to recovery, advice and education, functional-based exercise and pain.

SUMMARY:
This study aims to evaluate the whether receiving physiotherapy early after onset of the problem is better than waiting a few weeks to see if it gets better before starting physiotherapy. 80 people with sciatica will take part in the study, half of which will receive physiotherapy 2 weeks after seeing their G.P. The other half will receive physiotherapy at the usual time, around 6 weeks after seeing their G.P.

DETAILED DESCRIPTION:
Sciatica is a relatively common problem which is often caused by nerve compression or irritation due to a lower back (Lumbar) disc prolapse. The problem is likely to improve in time as the body heals itself. However, this can take many months or sometime years. Sciatica can be a very painful condition, it may cause pins and needles, numbness or weakness in the legs affected. This, can cause great difficulty for people carrying out normal day to day activities.

Physiotherapy is often used to help people with sciatica but in many places in the United Kingdom it can take many weeks or months to begin therapy.

This study aims to see if having physiotherapy at 2 weeks after the patient has seen their G.P helps them get back to normal day to day function. This will be compared with another group of patients who will have physiotherapy at the 'usual' time of around 6 weeks after they have seen their G.P.The investigators will also be interviewing participants for their views of sciatica and physiotherapy. Each patient will receive a goal orientated physiotherapy management programme with achievement of those goals acting as secondary outcomes. Primary outcomes are feasibility objectives including patient recruitment rates, acceptability of outcome measures and intervention and rates of adverse events.

This is a pilot study which means that the investigators won't be directly comparing the 2 groups, but seeing if doing a full-scale study in the future is going to be feasible.The investigators will do this by measuring several different things, such as whether patients want to take part in the study or not, whether the tests the investigators will perform are the right tests and to see if the patients and physiotherapists find the treatment useful.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18-70 years of age with unilateral LRS defined as pain and or sensory disturbance and or weakness in a dermatomal and or myotomal distribution.

Exclusion Criteria:

* Patients with bilateral LRS.
* Patients with 'red flag' signs and symptoms of potential serious pathology.
* Cancer at the time of the study.
* Proven vascular claudication.
* Cauda Equina Syndrome (CES).
* Spinal fracture within the last 3 months.
* Chronic regional pain syndromes.
* Recent lower limb fracture.
* CVA with physical or psychiatric disability.
* Poor English skills (necessitating the use of an interpreter and invalidating outcomes measures-ODI).
* Other significant co-morbidities preventing regular attendance at physiotherapy clinics.
* Patients with significant mental health problems for which treatment adherence may be difficult or psychologically disabling.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Ability to recruit patients | 26 weeks
  Ability to recruit patients within the 26 week limit
Patients willing to be randomised | 26 weeks
  The willingness of patients to be randomised will be collected together with reasons for not wanting to be randomised.
Ability to initiate treatment | 2 weeks for intervention arm, 6 weeks for control
  Demonstrate the ability to organise physiotherapy appointments expeditiously
Ensure patient safety | 52 weeks
  Record all adverse and serious adverse events

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | Baseline, 6 weeks, 12 weeks, 26 weeks
  self-rated disability 0/100
EQ5D-5L | Baseline, 6 weeks, 12 weeks, 26 weeks
  General health measurement
Back & leg pain | Baseline, 6 weeks, 12 weeks, 26 weeks
  Self-reported back and leg pain
Goal achievement | 26 weeks
  Patient will rate whether their goal(s) have been achieved

REFERENCES:
- [Derived] Reddington M, Walters SJ, Cohen J, Baxter SK, Cole A. Does early intervention improve outcomes in the physiotherapy management of lumbar radicular syndrome? Results of the POLAR pilot randomised controlled trial. BMJ Open. 2018 Jul 28;8(7):e021631. doi: 10.1136/bmjopen-2018-021631. PMID 30056385
- [Derived] Reddington M, Walters SJ, Cohen J, Baxter S. Does early intervention improve outcomes in physiotherapy management of lumbar radicular syndrome? A mixed-methods study protocol. BMJ Open. 2017 Mar 3;7(3):e014422. doi: 10.1136/bmjopen-2016-014422. PMID 28259854